CLINICAL TRIAL: NCT05940064
Title: Prospective Single-arm, Single-center Clinical Study of Zanubrutinib, Polatuzumab Vedotin and Rituximab (ZPR) Regimen in Elderly Treatment-naive Patients With Diffuse Large B-cell Lymphoma
Brief Title: Prospective Clinical Study of ZPR Regimen in Elderly Treatment-naive Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peng Liu (Other)
Responsible Party: Sponsor-Investigator, Peng Liu, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHZS-DLBCL003
Record Dates: First submitted 2023-06-19; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B Cell Lymphoma; Treatment-naive; Elderly; Zanubrutinib; Polatuzumab Vedotin; Rituximab; Efficacy; Safety
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; polatuzumab vedotin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly Treatment-naive Diffuse Large B-cell Lymphoma (Experimental): Elderly Treatment-naive Diffuse Large B-cell Lymphoma
  Interventions: Drug: Zanubrutinib, Polatuzumab Vedotin, Rituximab

INTERVENTIONS:
Drug: Zanubrutinib, Polatuzumab Vedotin, Rituximab — Drug: Zanubrutinib, Polatuzumab Vedotin and Rituximab Zanubrutinib（Z）160 mg bid po Day 1-21; Polatuzumab Vedotin（P）1.8 mg/kg ivgtt D1; Rituximab（R）375 mg/m^2 ivgtt D1
  Other Names: ZPR

SUMMARY:
This is a prospective, single-arm, single-center clinical study. This clinical study aims to explore the efficacy and safety of the ZPR（Zanubrutinib, Polatuzumab vedotin and Rituximab）regimen in elderly patients with treatment-naive diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center clinical study. This clinical study aims to explore the efficacy and safety of the ZPR（Zanubrutinib, Polatuzumab vedotin and Rituximab）regimen in elderly patients with treatment-naive diffuse large B-cell lymphoma.

Primary objective: use ORR to evaluate the efficacy of ZPR in treating elderly treatment-naive DLBCL patients

Secondary objective: Evaluate the safety of ZPR treatment for elderly treatment-naive DLBCL patients

The subjects received 6 cycles of ZPR regimen, one cycle every 21 days. Then Zanubrutinib alone will continue to be used until Zanubrutinib has been used for 1 year or disease progression or intolerable adverse effects, death, withdrawal of informed consent or study termination.

Zanubrutinib（Z）160 mg bid po Day 1-21; Polatuzumab vedotin（P）1.8 mg/kg ivgtt D1; Rituximab（R）375 mg/m^2 ivgtt D1.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled in this study:

1. Patients with histopathologically confirmed DLBCL;
2. Patients haven't received any anti-DLBCL therapy. Corticosteroids alone is not considered as a line of treatment;
3. The age of patients ≥ 70 years old, or between 60 and 69 but with an ECOG score between 2-4;
4. Patients intolerant to standard front-line therapy, i.e. R-CHOP, or R-miniCHOP etc.
5. Good organ function;
6. Measurable lesions detected by radiological imaging were defined as the longest diameter of at least 1 lymph node lesion > 1.5 cm, or the longest diameter of at least 1 extranodal lesion > 1.0 cm, and at least 2 vertical diameters that could be accurately measured;
7. Life expectancy ≥ 6 months;
8. Sign written informed consent.

Exclusion Criteria:

Patients with any of the following conditions cannot be enrolled in this study:

1. Patients with primary central nervous system lymphoma;
2. Patients with previous exposure to BTK inhibitors;
3. Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc; Currently clinically significant active cardiovascular disease, such as uncontrolled arrhythmia, congestive heart failure, any grade 3 or 4 heart disease defined by the New York Heart Association functional classification, or history of myocardial infarction within 6 months after screening. The left ventricular ejection fraction measured by echocardiography was < 50%;
4. Abnormal laboratory indicators at screening (unless caused by lymphoma):

   4.1 ANC<1.5×10^9/l, PLT<80×10^9/l 4.2 Coagulation function: INR greater than 1.5 times the upper limit of normal value; Pt and APTT were greater than 1.5 times the upper limit of normal 4.3 Liver function: ALT or ast was 2 times higher than the upper limit of normal, AKP and bilirubin were 1.5 times higher than the upper limit of normal 4.4 Renal function: creatinine was 1.5 times higher than the upper limit of normal, creatinine clearance rate was < 60 ml/min (estimated according to Cockcroft Gault formula)
5. HIV-infected persons;
6. HCV active infection;
7. HBsAg positive patients need to be HBV DNA negative before enrollment; In addition, if the patient is HBsAg negative but HBcAb positive (regardless of HBsAb status), HBV DNA testing is still required. If the result is positive, antiviral treatment is required, and HBV DNA is required to be negative before enrollment;
8. Other concurrent and uncontrolled medical conditions that the investigator believes will affect the patient's participation in the study, including psychiatric patients or other patients who are known or suspected to be unable to fully comply with the study protocol;
9. Known allergy to test drug;
10. Inability to swallow capsules or suffering from diseases that seriously affect gastrointestinal function, such as malabsorption syndrome, gastrectomy or small bowel resection, symptomatic inflammatory bowel disease, or partial or complete intestinal obstruction;
11. Pregnant or lactating women;
12. Corticosteroids (dose equivalent to prednisone > 20 mg/ day) were previously given for antitumor purposes within 7 days, and chemotherapy, targeted therapy, or radiotherapy were previously received within 3 weeks, or antibody-based therapy was received within 3 weeks, or traditional Chinese medicine anticancer therapy was performed within 4 weeks;
13. Major surgery was performed within 4 weeks after screening;
14. Sustained treatment with potent and moderate CYP3A inhibitors or CYP3A inducers is needed. Patients could not be enrolled if they had taken potent and moderate CYP3A inhibitors or CYP3A inducers within 7 days before the first administration of study drugs (or had taken these drugs for no more than 5 half-lives).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR at the end of the 6th treatment cycle | about six months from the start of ZPR
  the proportion of participants who have achieved complete or partial remission determined by the researcher.

SECONDARY OUTCOMES:
CRR at the end of the 6th treatment cycle | about six months from the start of ZPR
  the proportion of subjects evaluated by researchers to obtain CR.
Proportion of patients who have achieved 2-year PFS | 2-year (from the start of treatment to the first recording of disease progression or death, based on the investigator's assessment of the first occurrence)
  Defined as the proportion of participants with a time of 2 years from the start of treatment to the first recording of disease progression or death, based on the investigator's assessment of the first occurrence
Safety evaluation | between the first administration of the study drug and 30 days after discontinuation, or during the progression of the disease or the initiation of new anticancer treatment, whichever came first
  incidence and severity of adverse events (AE) and Serious adverse event (SAE) during the study

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, Ph.D, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No